CLINICAL TRIAL: NCT01113580
Title: A Phase IV, Single-centre, Open-label Study to Evaluate the Immunogenicity and Safety of the 2010/2011 Formulation of Enzira® Vaccine in Two Groups of Healthy Volunteers: 'Adults' (Aged 18 to 59 Years) and 'Older Adults' (Aged 60 Years or Older)
Brief Title: A Clinical Trial of CSL's 2010/2011 Formulation of Enzira® in a Healthy Adult Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-ASU-10-66; 2010-019532-12 (EudraCT Number)
Record Dates: First submitted 2010-04-26; First posted 2010-04-30 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adults (Experimental): Healthy volunteers aged 18 to 59 years
  Interventions: Biological: CSL's 2010/2011 Formulation of Enzira® Vaccine
- Older Adults (Experimental): Healthy volunteers aged 60 years or older
  Interventions: Biological: CSL's 2010/2011 Formulation of Enzira® Vaccine

INTERVENTIONS:
Biological: CSL's 2010/2011 Formulation of Enzira® Vaccine — 45 mcg of HA antigen in 0.5 mL administered by intramuscular injection into the deltoid region of the arm on Day 0

SUMMARY:
The purpose of this study is to determine whether the 2010/2011 Formulation Enzira vaccine is safe and elicits an immune response to seasonal influenza in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and older at the time of the first study vaccination.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza virus vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of the Study Vaccine.
* Clinical signs of an active infection
* Vaccination with a seasonal or experimental influenza virus vaccine in the 6 months preceding study entry
* Females who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Beboso, Dr, Principal Investigator — Chiltern (Early Phase) Limited
Locations (1):
- Chiltern (Early Phase) Limited, Dundee, Angus and Dundee, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adults | Older Adults
Started | 60 | 60
Completed | 59 | 60
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults | Older Adults | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0
  18 to 59 years | 60 | 0 | 60
  >= 60 years | 0 | 60 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 31 | 36 | 67

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Evaluable Participants Achieving Seroconversion or Significant Increase in Antibody Titre.
Description: As per the criteria specified in the CPMP/BWP/214/96 Note for Guidance on Harmonisation of Requirements for Influenza Vaccines. For haemagglutination inhibition (HI), seroconversion is defined as achieving a post-vaccination titre of ≥ 40 for those participants with a pre-vaccination HI titre of < 10; significant increase is defined as a four-fold or greater increase in HI titre for those participants with a pre-vaccination HI titre of ≥ 10.
Time Frame: Approximately 21 days after vaccination
Population: The Evaluable Population comprised all participants who were vaccinated with the study vaccine, provided both pre- and post-vaccination antibody titre results, and were not excluded from the analyses (eg, for the use of a prohibited medication or a laboratory-confirmed influenza virus infection between Visits 1 and 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 58 | 60
Percentage of participants
  A/California/7/2009 (H1N1)-like strain | 89.7 [78.8 to 96.1] | 80.0 [67.7 to 89.2]
  A/Perth/16/2009 (H3N2)-like strain | 89.7 [78.8 to 96.1] | 71.7 [58.6 to 82.5]
  B/Brisbane/60/2008-like strain | 63.8 [50.1 to 76.0] | 28.3 [17.5 to 41.4]

2. Primary Outcome: The Geometric Mean Fold Increase (GMFI) in Antibody Titre After Vaccination.
Description: GMFI is defined as the geometric mean of the fold increases of post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Fold increase
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 58 | 60
Fold increase
  A/California/7/2009 (H1N1)-like strain | 20.48 [14.714 to 28.512] | 12.90 [8.218 to 20.239]
  A/Perth/16/2009 (H3N2)-like strain | 24.70 [16.967 to 35.958] | 11.53 [7.313 to 18.191]
  B/Brisbane/60/2008-like strain | 6.63 [4.598 to 9.571] | 2.77 [2.055 to 3.747]

3. Primary Outcome: The Percentage of Evaluable Participants Achieving a HI Titre ≥ 40 or Single Radial Haemolysis (SRH) Area ≥ 25 mm2.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 58 | 60
Percentage of participants
  A/California/7/2009 (H1N1)-like strain | 91.4 [81.0 to 97.1] | 90.0 [79.5 to 96.2]
  A/Perth/16/2009 (H3N2)-like strain | 98.3 [90.8 to 100.0] | 96.7 [88.5 to 99.6]
  B/Brisbane/60/2008-like strain | 89.7 [78.8 to 96.1] | 70.0 [56.8 to 81.2]

4. Secondary Outcome: Frequency of Any Solicited Adverse Events (AEs)
Description: The number of participants reporting any solicited AEs.
Time Frame: During the 4 days after vaccination (Day 0 plus 3 days)
Population: The Safety Population comprised all participants who received study vaccine and provided follow-up safety data.
Measure: Number; unit: participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
participants
  Any local solicited AE | 32 | 18
  Any induration larger than 50 mm | 2 | 0
  Any erythema | 22 | 9
  Any ecchymosis | 5 | 4
  Any pain | 22 | 10
  Any general (systemic) solicited AE | 4 | 3
  Any temperature above 38 degrees C for ≥ 24 hours | 0 | 3
  Any chills | 4 | 2
  Any malaise | 3 | 2

5. Secondary Outcome: Frequency and Intensity of Any Unsolicited Adverse Events
Description: Unsolicited adverse event (UAE) grading:
  Mild: Symptoms were easily tolerated and there was no interference with daily activities. Moderate: Enough discomfort to have caused some interference with daily activities. Severe: Symptoms that prevented normal, everyday activities.
Time Frame: After vaccination until the end of the study; approximately 21 days
Population: The Safety Population comprised all participants who received study vaccine and provided follow-up safety data.
Measure: Number; unit: participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
participants
  Number of participants with at least one UAE | 28 | 22
  Number of participants reporting mild UAE | 22 | 19
  Number of participants reporting moderate UAE | 7 | 2
  Number of participants reporting severe UAE | 3 | 2

ADVERSE EVENTS:
Time Frame: Approximately 21 days after study vaccination for serious adverse events and unsolicited adverse events.
Description: Other adverse events presented were unsolicited adverse events up to approximately 21 days after study vaccination.
Arm/Group | Adults | Older Adults
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 22/60 | 15/60
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (N=60) | Older Adults (N=60)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 12 (12) | 4 (4)
Influenza like illness (General disorders) | 3 (3) | 2 (2)
Vaccination site erythema (General disorders) | 2 (2) | 1 (1)
Vaccination site induration (General disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.